CLINICAL TRIAL: NCT05293262
Title: Definitive Endourological Interventions for Urolithiasis Management During COVID19- Outcomes From a Cohort Study
Brief Title: Endourological Management of Stones During COVID19
Status: Completed | Type: Observational
Sponsor: Roxanne Teo (Other)
Responsible Party: Sponsor-Investigator, Roxanne Teo, Medical Officer, National University Health System, Singapore
Organization: National University Health System, Singapore (Other)
Other Study IDs: 2020/01298
Record Dates: First submitted 2022-03-13; First posted 2022-03-24 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Urolithiasis; COVID-19
Keywords: endourology; pandemic
MeSH Terms: conditions — Urolithiasis; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who underwent endourological surgery for urolithiasis during COVID19: Endourological surgery (including ureteral stent insertion, ureteroscopy, retrograde intrarenal surgery)
  Interventions: Procedure: Endourological surgery

INTERVENTIONS:
Procedure: Endourological surgery — Includes ureteral stent insertion, ureteroscopies and retrograde intrarenal surgeies

SUMMARY:
Guidelines for endourological procedures during COVID-19 have suggested deferring all elective procedures, while obstructed/ infected stones should undergo urgent decompression.

At our centre, screening protocols were implemented with prioritization strategies so that elective care could safely continue at deescalated rates. COVID or septic patients underwent emergency decompression, while non-COVID and non-septic patients underwent primary ureteroscopy (URS) or retrograde intrarenal surgery (RIRS).

We aim to report our experience with endourological surgery for stone disease during COVID-19.

DETAILED DESCRIPTION:
We conducted a retrospective review of a prospectively maintained database of all endourological surgeries for stones in our centre during the first wave of COVID19.

ELIGIBILITY:
Inclusion criteria

- all patient with urolithiasis who underwent endourological interventions during COVID19 pandemic

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with obstructing urolithiasis who underwent decompression of ureteric stents, ureteroscopy or retrograde intrarenal surgery with laser lithotripsy during the period of study in our institution were included in the study
Sampling Method: Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2020-01-23 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Length of hospital stay | From admission to discharge from hospital, up to 3 months
  Length of hospital stay
Complication rate | From admission up to 3 months post operatively
  Complications as defined by Clavien Dindo classification system
Stone free rate | At follow up visit in clinic 3 months post procedure

SECONDARY OUTCOMES:
Readmission rate | From discharge up to three months post operatively

CONTACTS AND LOCATIONS:
Overall Officials: Chin Tiong Heng, Principal Investigator — Ng Teng Fong General Hospital
Locations (1):
- Ng Teng Fong General Hospital, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No